CLINICAL TRIAL: NCT03844399
Title: Use of 3-Dimensional (3D) Ultrasound Imaging to Guide the Treatment of Abdominal Tumours Using Focal Ablation or Biopsies
Brief Title: (3D) Ultrasound Imaging Liver and Kidney
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 6319
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-07

CONDITIONS: Liver Cancer; Kidney Cancer
Keywords: Diagnostic; Intervention; 3D Ultrasound
MeSH Terms: conditions — Liver Neoplasms; Kidney Neoplasms; Disease | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Cancer patients who are scheduled to undergo an ablation or biopsy of a liver or kidney tumour
  Interventions: Device: Ablation; Device: Biopsy

INTERVENTIONS:
Device: Ablation — The medical device will passively record image data during the standard care ablation
Device: Biopsy — The medical device will passively record image data during the standard care biopsy

SUMMARY:
This study is to assess the addition of 3D ultrasound guidance during standard care ablation or biopsies of liver or kidney tumours. 3D ultrasound only differs from conventional 2D ultrasound in that the ultrasound transducer is mounted on a special assembly that moves the transducer in precise, stepped movements while a succession of 2D images are collected by the computer. Special software written specifically for 3D ultrasound precisely aligns these 2D images into a 3-demensional volume , allowing area in question to be viewed in many different planes. 3D ultrasound is a safe, fast, non-invasive imaging procedure. Ultrasound images will be checked against the pre- and post- procedure CT images to make sure the tumours were completely removed or properly targeted during biopsy.

DETAILED DESCRIPTION:
Images will be acquired by a physician on patients who are undergoing a liver or kidney ablation or biopsy procedure who are well enough to provide consent. Patients will be imaged during the ablation procedure according to the standard of care, and subsequent analysis will commence following the acquisition. The devices being used are all property of the LHSC health network that have been licensed for clinical use through Health Canada. In addition, 3D ultrasound only differs from conventional 2D ultrasound in that the ultrasound transducer is mounted on a special assembly that moves the transducer in precise, stepped movements while a succession of 2D images are collected by the computer. Special software written specifically for 3D ultrasound precisely aligns these 2D images into a 3-dimensional volume, allowing the area in question to be viewed in different planes. The clinical 2D an d3D ultrasound images will be checked against the pre- and post- procedure CT images to make sure the tumours were completely removed.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are scheduled for standard care liver or kidney ablation or biopsy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion / exclusion criteria, who are already scheduled for a liver or kidney tumour ablation or biopsy will be selected for the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Needle Guidance Intervention | April 2020
  The objective of this study is to use 3D ultrasound in addition to standard care ultrasound to guide the ablation needles in destroying focal tumours within the diseased organ

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada